CLINICAL TRIAL: NCT03737409
Title: PFOX: Pulmonary Fibrosis Ambulatory Oxygen Trial
Acronym: PFOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Anne E Holland PhD, FThorSoc, Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC/18/Alfred/42
Record Dates: First submitted 2018-09-18; First posted 2018-11-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Fibrotic Interstitial Lung Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen therapy with POC (AOT group) (Experimental): Patients will receive ambulatory oxygen therapy provided by a portable oxygen concentrator and will be encouraged to use it at all times when they are moving about, including walking at home or in the community, during exercise or during other activities.
  Interventions: Other: Ambulatory Oxygen Therapy
- Sham oxygen therapy with POC (air group) (Sham Comparator): Patients will receive sham ambulatory oxygen therapy provided by a portable oxygen concentrator and will be encouraged to use it at all times when they are moving about, including walking at home or in the community, during exercise or during other activities.
  Interventions: Other: Sham Ambulatory Oxygen Therapy

INTERVENTIONS:
Other: Ambulatory Oxygen Therapy — Supplemental oxygen delivered during exercise and activities of daily living via a portable oxygen concentrator
  Arms: Oxygen therapy with POC (AOT group)
Other: Sham Ambulatory Oxygen Therapy — Air delivered during exercise and activities of daily living via a portable oxygen concentrator that has been modified to deliver air
  Arms: Sham oxygen therapy with POC (air group)

SUMMARY:
The fibrotic interstitial lung diseases (fILD) are characterised by lung scarring, distressing breathlessness and poor health-related quality of life. Exertional desaturation (low blood oxygen during exercise) is a hallmark of fILD, occurring in over 50% of patients. It is sometimes treated with ambulatory oxygen therapy (AOT), which involves breathing supplemental oxygen during physical activity. However the absence of clinical trials has given rise to marked variations in policy and practice globally. Even where AOT is available, treatment adherence using the traditional delivery method of cylinder gas is poor. Recently new devices called portable oxygen concentrators (POCs), have become available, which are lighter and more maneuverable than a cylinder. This may enhance adherence and maximize treatment benefits.

This trial will determine the clinical benefits and societal costs of AOT for people with fILD and exertional desaturation. A randomised controlled trial with blinding of participants, assessors and clinicians, and an embedded economic evaluation will be conducted. A total of 260 participants with fILD and exertional desaturation will be randomly assigned to use either AOT or air delivered using a POC for 6 months. If this trial demonstrates clinical and economic benefits of AOT then the findings can be rapidly translated into practice.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILDs) are characterized by scarring of lung tissue. Stiffening of the lungs leads to reduced transfer of oxygen into the blood, decreased exercise capacity and premature death. Around 85% of the ILDs are known as fibrotic ILD (fILD), a form of ILD which tends to have worse outcomes than other types of ILD. People with fibrotic ILD often experience distressing breathlessness, cough and fatigue; loss of independence and life roles; financial strain; and unpleasant treatment side effects.The most common of the fILDs is idiopathic pulmonary fibrosis (IPF), which has an average survival of 3 years from diagnosis. Recently, two new treatments have been shown to halve the annual decline in lung function in mild to moderate IPF, making it a 'treatable' condition for the first time. However, these treatments only slow the decline in lung function; they do not stabilize or reverse it, nor do patients experience improved quality of life or breathlessness.

For people with fILD who have abnormally low oxygen in the blood at rest, long term oxygen therapy (LTOT, used ≥18 hours per day) is strongly recommended, based on survival benefits in studies of people with chronic obstructive pulmonary disease (COPD). However, for people with fILD who have low oxygen levels only during exertion, the role of oxygen therapy is not clear.

Ambulatory oxygen therapy (AOT), defined as the use of oxygen during exercise and activities of daily living, has historically been used to improve blood oxygen levels and exercise capacity. However, many people with fILD find this treatment difficult to use. Oxygen cylinders are heavy and run out quickly, therefore patient burden often exceeds any benefits. Portable oxygen concentrators (POCs) are newly available, lighter and rechargeable. However there are potential disadvantages to POCs. Generally, they deliver oxygen in pulses, which is where oxygen is delivered only when breathing in, and they do not deliver 100% oxygen. Doctors often express concerns that POCs cannot meet the demands of people with fILD during exercise. Recently it was shown that people with fILD who use a POC have similar blood oxygen levels to those who use a cylinder during exercise, suggesting that this might be a useful treatment.

This study will examine the benefits and costs of ambulatory oxygen, delivered using a POC, in people with fILD and exertional desaturation. The aim is to compare the impact of AOT vs air in people with fILD who have low blood oxygen during exercise, and to compare the cost-effectiveness of AOT and air in fILD. A total of 260 people with fILD will be invited to participate. The trial will be conducted at four sites in Australia and two sites in Sweden. Participants will be randomly allocated into two groups; Group 1 will be administered AOT using a POC (AOT group); and Group 2 will be administered sham AOT using an identical POC (air group). Participants, health professionals and trial staff will not be aware of which POC is being used. The allocated treatment will be delivered for 6 months. Measurements of physical activity during daily life, symptoms, exercise capacity and HRQOL will be collected at the beginning of the trial, and 3 and 6 months after treatment has commenced. Information about use of health care services, both from hospital records and directly from participants will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Fibrotic Interstitial Lung Disease
* Stable pharmacotherapy over the last 3 months
* Exertional desaturation (SpO2≤88% for at least 10 consecutive seconds) during a 6 Minute Walking Test performed on room air

Exclusion Criteria:

* Currently using or eligible for long term oxygen therapy (PaO2≤55 mmHg at rest on room air, or 56-59 mmHg with evidence of right heart failure)
* Current smokers
* Pregnant patients
* Patients cognitively unable to consent; or if death or transplant is anticipated within the study period.
* Participants currently in pulmonary rehabilitation
* Non-ambulant patients
* Admission to an acute care hospital within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity measured by steps per day | Baseline, 3 month and 6 month assessments
  Steps per day assessed by activity monitors

SECONDARY OUTCOMES:
Change in functional exercise capacity assessed by 6-minute walk distance | Baseline, 3 month and 6 month assessments
  Distance in meters achieved on a 6-minute walk test
Change in health related quality of life evaluated using the St George's Respiratory Questionnaire | Baseline, 3 month and 6 month assessments
  St George's Respiratory Questionnaire is a disease-specific health related quality of life questionnaire.The questionnaire is divided in 3 domains: Symptoms (frequency and severity), Activity (activities that cause or are limited by breathlessness) and Impact (social functioning and psychological disturbances resulting from airways disease). Values of each domain as well as the total score value will be reported. Each item is weighted based on empirical data. Total score and scores in each domain can range from 0 to 100. Higher scores indicate more limitations in quality of life.
Change in dyspnea measured using the Dyspnea-12 questionnaire | Baseline, 3 month and 6 month assessments
  Dyspnea-12 is a uni-dimensional 12-item questionnaire divided in 2 domains: physical items (1 to 7) and affective items (8-12). Each item evaluate breathing experience and can be scored as: None (0), Mild (1), Moderate (2) or Severe (3). Results of this questionnaire will be reported as total score that can range from 0 to 36 and separate scores that can range from 0 to 21 for physical component and 0 to 15 for affective component. Higher scores indicate worse dyspnea.
Changes in fatigue evaluated by the Fatigue Severity Scale | Baseline, 3 month and 6 month assessments
  Fatigue Severity Scale (FSS), a self reported rating scale including 9 items to measure how fatigue affects motivation, exercise, physical functioning, carrying out duties and how fatigue interferes with work, family, or social life. Each item is scored on a 7 point scale in which 1 = strongly disagree and 7= strongly agree. Total score range from 9 to 63. Higher scores indicate greater fatigue severity.
Change in anxiety and depression measured by the Hospital Anxiety and Depression Scale | Baseline, 3 month and 6 month assessments
  Hospital Anxiety and Depression Scale (HADS), a scale with 14 items divided into two domains : anxiety symptoms (7 items) and depression symptoms (7 items). Each item can be scored from 0 to 3. Scores from each domain can vary from 0 to 21 and are stratified as follows: 0-7 (indicates absence of anxiety/depression symptoms); 8-10 ( presence of symptoms of anxiety and depression in moderate degree - borderline); 11 or more (significant number of anxiety/depression symptoms - confirmed cases). Score of each domain as well as number of confirmed cases will be reported.
Change in time spent in moderate to vigorous physical activity | Baseline assessment, 3 month and 6 month assessments
  Time spent in moderate to vigorous physical activity, measured by a wrist-worn, tri-axial accelerometer.
Change in sedentary time | Baseline assessment, 3 month and 6 month assessments
  Time spent sedentary, measured by a wrist-worn, tri-axial accelerometer.
Skeletal muscle metabolism | Baseline, 3 month and 6 month assessments
  Plasma markers of skeletal muscle metabolism (xanthine, hypoxanthine [units pmole/µL]) will be analysed from collected blood samples.
Systemic inflammation | Baseline, 3 month and 6 month assessments
  C-reactive protein [unit ng/mL]) will be analysed from collected blood samples.
Oxidative stress | Baseline, 3 month and 6 month assessments
  Thiobarbituric acid reactive substrates [units µM]) will be analysed from collected blood samples.
Use of oxygen therapy | 3 month and 6 month assessments
  Hours of usage of the portable concentrator.
Oxygen saturation in daily life | 3 month and 6 month assessments
  Wrist oximeter that will be worn during waking hours on two consecutive weekdays.
Incremental cost-effectiveness ratio | 6 month assessment
  Difference in health care costs compared to differences in quality-adjusted life years -QALYs

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holland, Professor, Principal Investigator — Monash University
Locations (1):
- Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after deidentification of participants after publication, with approval of the Alfred Health Human Research Ethics Committee.
Supporting Information: Study Protocol
Time Frame: 9-36 months after article publication
Access Criteria: Proposals submitted to corresponding author and approved by Alfred Hospital Human Research Ethics Committee.

REFERENCES:
- [Derived] Kawachi S, Hoffman M, Holland AE. Clinical Features Associated With Fatigue in People With Fibrotic Interstitial Lung Disease: Cross-Sectional Study. Respirology. 2025 Nov;30(11):1087-1093. doi: 10.1111/resp.70091. Epub 2025 Jul 20. PMID 40685600
- [Derived] Hoffman M, Burge AT, Wong N, McDonald CF, Chambers DC, Glaspole I, Mackintosh JA, Ekstrom M, Skold M, Goh NSL, Corte TJ, Holland AE. Exertional Desaturation During the 6-Minute Walk Test vs Daily Life in People With Fibrotic Interstitial Lung Disease. Chest. 2024 Mar;165(3):632-635. doi: 10.1016/j.chest.2023.08.024. Epub 2023 Sep 1. No abstract available. PMID 37659620
- [Derived] Holland AE, Corte T, Chambers DC, Palmer AJ, Ekstrom MP, Glaspole I, Goh NSL, Hepworth G, Khor YH, Hoffman M, Vlahos R, Skold M, Dowman L, Troy LK, Prasad JD, Walsh J, McDonald CF. Ambulatory oxygen for treatment of exertional hypoxaemia in pulmonary fibrosis (PFOX trial): a randomised controlled trial. BMJ Open. 2020 Dec 13;10(12):e040798. doi: 10.1136/bmjopen-2020-040798. PMID 33318119

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03737409/SAP_000.pdf